CLINICAL TRIAL: NCT04250324
Title: A Phase I Clinical Study of CD19-targeted Chimeric Antigen Receptor (CAR) T Cells Injection, for Relapsed and Refractory (R/R) Large B-cell Lymphoma
Brief Title: Study of Safety and Efficacy of BZ019 in (R/R) Large B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XY2019028-EC-1
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Large B-cell Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BZ019 (Experimental): The subjects are enrolled into 2 dose-escalation cohorts, include 3x10^6/kg、6x10^6/kg, and dose-expansion cohorts, maybe 8x10^6/kg、10x10^6/kg.
  Interventions: Biological: BZ019

INTERVENTIONS:
Biological: BZ019 — A treatment program will include lymphodepleting chemotherapy with fludarabine and cyclophosphamide (flu/cy) followed by single-dose of BZ019 administered intravenously (IV).

SUMMARY:
This is an open-label, multicenter, dose-escalation phase 1 study to determine the Safety and Efficacy of BZ019 in relapsed or refractory CD19+ B-cell Lymphoma subjects.

DETAILED DESCRIPTION:
This is an open-label, multicenter, phase 1 study to determine the safety, PK, and antitumor activity of BZ019 in adult subjects with R/R large CD19+B cell lymphoma. The safety and efficacy of a single dose of different target doses of BZ019 will be evaluated in the dose-escalation phase and dose-expansion phase.

Primary objectives:

- To evaluate the safety and tolerance of single infusion of BZ019 in adult patients with relapsed or refractory large B-cell lymphoma, and to determine the maximum tolerable dose (MTD) and phase II recommended dose.

Secondary objectives：

* To evaluate the pharmacokinetics and survival of BZ019 in the peripheral blood of adult patients with relapsed or refractory large B-cell lymphoma;
* To evaluate the Pharmacodynamic characteristics of BZ019 in adult patients with relapsed or refractory large B-cell lymphoma;
* Objective response rate (ORR), Overall survival, progression free survival, event free survival, and tumor progression time were used to evaluate the antitumor efficacy of BZ019 in the treatment of relapsed or refractory large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures;
* Age ≥ 18 years subjects with Relapsed or refractory large B-cell lymphoma, only DLBCL non-specific type, primary mediastinal large B-cell lymphoma, follicular lymphoma transformed large B-cell lymphoma, advanced B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement, advanced B-cell lymphoma non-specific type. The definition of refractory is as follows:

  * no response to the last treatment, including:The best response to the latest treatment is disease progression (PD), or the best response to the latest treatment plan is disease stability (SD) and the maintenance time is not more than 6 months after the last administration;
  * or not suitable for autologous hematopoietic stem cell transplantation (ASCT), or ASCT refractory, including: disease progression after ASCT or recurrence within ≤ 12 months (recurrence must be confirmed by biopsy), or if receiving remedial treatment after ASCT, the subject must have no reaction or recurrence after the last treatment.
* Subjects must be accepted adequate treatment before and have received at least 2 lines of treatment or relapse or progress after autologous hematopoietic stem cell transplantation, and the treatment history at least include:

  * Treatment by CD20 monoclonal antibody (Rituximab) except for CD20 negative;
  * a chemotherapy regimen containing anthracyclines.
* According to the preliminary evaluation, staging and response evaluation recommendations for Hodgkin and non Hodgkin's lymphoma (2014 Edition), at least one measurable lesion was found in the screening period.
* Life expectancy ≥12 weeks.
* Baseline Eastern Cooperative Oncology Group (ECOG) score is 0 or 1 .
* Adequate organ function:

  * Renal function defined as:A serum creatinine of ≤1.5 x ULN or Estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/min/1.73 m^2;
  * Liver function defined as:Alanine Aminotransferase (ALT) ≤ 5 x ULN；Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert-Meulengracht syndrome; patients with Gilbert-Meulengracht syndrome may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN;
  * Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation > 91% on room air.
* Hemodynamically stable and Left Ventricle Ejection Fraction (LVEF) ≥ 50%, confirmed by echocardiogram or Multigated Radionuclide Angiography (MUGA).
* No blood transfusion within 1 week before signing the informed consent, sufficient bone marrow reserve is available, which is defined as:

  * Absolute neutrophil count (ANC) > 1000/μl;
  * Absolute lymphocyte count (ALC) ≥ 500/μl;
  * Platelets ≥ 50000/μl;
  * Hemoglobin > 8.0 g/dl, for patients with bone marrow invasion, hemoglobin > 6.0 g/dl can be considered into the group.
* Must have an apheresis product of non-mobilized cells accepted for manufacturing.
* If the patient uses the following drugs, the following conditions should be met:

  * glucocorticoids: The treatment dose of glucocorticoids must be stopped 72 hours before BZ019 infusion. However, glucocorticoids of physiological alternative dose are allowed: prednisone or its equivalent ≤ 15 mg / day;
  * Immunosuppression: Any immunosuppressive medication must be stopped ≥ 4 weeks prior to enrollment;
  * Antiproliferative therapies other than lymphodepleting chemotherapy within two weeks of infusion
  * Antibody use including anti-CD20 therapy within 4 weeks prior to infusion or 5 half-lives of the respected antibody, whichever is longer
  * CNS disease prophylaxis must be stopped > 1 week prior to BZ019 infusion (e.g. intrathecal methotrexate)
* Women of child-bearing age and all male subjects must agree to use effective contraceptive methods until BZ019 are no longer present in the body (detected by PCR).

Exclusion Criteria:

* Patients who have previously received any anti-CD45, anti-CD19 or anti-CD3 therapy;
* Patients who have previously received any adoptive T cell therapy or gene therapy products, including CAR-T therapy;
* Active Central Nervous System (CNS) involvement by malignancy or secondary CNS involvement
* History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or self-immune disease with CNS involvement.
* Prior allogeneic HSCT.
* Chemotherapy other than lymphodepleting chemotherapy within 2 weeks of infusion.
* Investigational medicinal product within the last 30 days prior to screening.
* Prior radiation therapy within 6 weeks of infusion.
* Patients with positive hepatitis B (HBsAg and / or HBcAb positive, except for those with positive surface antibody alone) or hepatitis C serological markers;
* HIV positive or Treponema pallidum positive patients.
* Patients with uncontrollable active or life-threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours before infusion);
* Patients with unstable angina and / or myocardial infarction within 6 months before screening, or patients with serious or uncontrollable other diseases (such as unstable or uncompensated respiratory, heart, liver or kidney diseases) during screening;
* Previous or concurrent malignancy with the following exceptions:

  * Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
  * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to the study
  * A primary malignancy which has been completely resected and in complete remission for ≥ 5 years
* Pregnant or nursing (lactating) women.
* Patients with uncontrolled arrhythmia.
* Patients on oral anticoagulation therapy within 1 week prior to BZ019 infusion.
* Patients with active neurological auto immune or inflammatory disorders(e.g. Guillain Barre Syndrome, Amyptrophic Lateral Sclerosis)
* Other protocol-related inclusion/exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | After 28 days of single infusion
  Safety
Maximum tolerated dose (MTD) | After 28 days of single infusion
  Tolerability

SECONDARY OUTCOMES:
Pharmacokinetics（the copies of cells in vivo） | Month 24
  Pharmacokinetics is defined as the number of copies of BZ019 DNA in peripheral blood at each visit after infusion until the test results are negative or below the detection limit. It aims to calculate the Peak Plasma Concentration (Cmax)
Pharmacokinetics（the duration of survival of cells in vivo） | Month 24
  Duration of BZ019 persistence is the period from the day of infusion to the first negative test result. It aims to calculate the area under the plasma concentration versus time curve (AUC)
Pharmacodynamics | After 28 days of single infusion
  Pharmacodynamics is defined as the level of Cytokine, at least include IL-2, IL-4, IL-6, IL-10, IL-15, IFN-γ, TNF-α. The peak value of cytokines and their return to baseline were evaluated
Antitumor efficacy-Objective response rate (ORR) | Month 24
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%)
Antitumor efficacy-Overall survival (OS) | Month 24
  The period from the first infusion to any cause of death
Antitumor efficacy-Progression-free survival (PFS) | Month 24
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first.
Antitumor efficacy-event -free survival (EFS) | Month 24
  Event free survival rate refers to the time from enrollment to occurrence of any event, including death, disease progression, change of chemotherapy program, change to chemotherapy, additional treatment, occurrence of lethal or intolerable side effects and other events.
Antitumor efficacy- Tumor progression time (TTP) | Month 24
  Tumor progression time refers to the time from the beginning of the infusion of cells to tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Ph.D, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin
  - Tianjin medical university cancer institute and hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No